CLINICAL TRIAL: NCT00527215
Title: A Study of Darbepoetin Alfa Administered Once Every Four Weeks in Chronic Renal Insufficiency (CRI) Subjects With Anemia
Brief Title: Phase 2 Study of Darbepoetin Alfa Extended Dosing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20010212
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2009-05-22 (Estimated); Status verified 2009-05

CONDITIONS: Pre-Dialysis
MeSH Terms: interventions — Darbepoetin alfa

ARMS (1):
- darbepoetin alfa (Experimental)
  Interventions: Drug: darbepoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa — starting dose determined by calculating a subject's total dose in the month preceding enrollment. Administered QM for 25 weeks. Change made as necessary to maintain a hemoglobin concentration within the target range os 10.0 - 12.0 g.dL

SUMMARY:
Multicenter, open label single arm study in which 140 subjects with CRI who are currently receiving SC darbepoetin alfa once every other week will receive darbepoetin alfa once every 4 weeks for 24 weeks. Upon enrollment into this study, subjects will receive darbepoetin alfa once every 4 weeks for 24 weeks. The initial dose will be equivalent to the subject's total dose in the month preceding enrollment. Doses may be titrated to maintain the Hb concentration in the target range.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* CRI with a creatinine clearance of greater than 15 but less than 40 mL/min
* Stable once every other week darbepoetin alfa SC for at least 6 weeks
* Hb values during screening / baseline of 10.0 - 12.0 g/dL
* Serum B12 and folate levels above the lower limit of normal and iron replete

Exclusion Criteria:

* Receiving renal replacement therapy
* Uncontrolled hypertension
* Hyperparathyroidism
* Major surgery, active inflammatory disease, receiving antibiotics, HIV-positive
* Current malignancy
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2002-03; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
To assess the proportion of CRI subjects maintaining a target hemoglobin (Hb) range of 10.0 to 12.0 g/dL when administered subcutaneous (SC) darbepoetin alfa once every 4 weeks | Study weeks 21 - 29

SECONDARY OUTCOMES:
To assess the safety, toleratbility, and pharmacokinetic (PK) profile of darbepoetin alfa when administered once every 4 weeks. | Entire study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Ling B, Walczyk M, Agarwal A, Carroll W, Liu W, Brenner R. Darbepoetin alfa administered once monthly maintains hemoglobin concentrations in patients with chronic kidney disease. Clin Nephrol. 2005 May;63(5):327-34. doi: 10.5414/cnp63327. PMID 15909591
- [Result] Agarwal A, Silver MR, Walczyk M, Liu W, Audhya P. Once-monthly darbepoetin alfa for maintaining hemoglobin levels in older patients with chronic kidney disease. J Am Med Dir Assoc. 2007 Feb;8(2):83-90. doi: 10.1016/j.jamda.2006.07.007. Epub 2006 Sep 29. PMID 17289537
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_33_NESP_20010212.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com